CLINICAL TRIAL: NCT00740428
Title: The Effectiveness of Pelvic Floor Exercises During Gestation in the Prevention of Urinary Incontinence and Pelvic Floor Muscle Dysfunction.
Brief Title: Pelvic Floor Exercises During Gestation in the Prevention of Urinary Incontinence and Pelvic Floor Muscle Dysfunction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: São Paulo State Health Department (Unknown); Assis Health Secretariat (Unknown)
Responsible Party: Adriano Dias, Botucatu Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: upeclin/HC/FMB-Unesp-10
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Pelvic Floor Abnormalities
Keywords: Pelvic floor,; muscular dysfunction,; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- G1 (Experimental): pregnants for the first time who will receive the physical therapy guide
  Interventions: Procedure: Pregnants for receive the physical therapy guide

INTERVENTIONS:
Procedure: Pregnants for receive the physical therapy guide — pregnants for the first time who will receive the physical therapy guide, perform the exercises under the supervision of a physical therapist, and complete an exercise compliance form and a log with information on urinary losses.
  Other Names: Physical therapy guide

SUMMARY:
Urinary incontinence is any involuntary loss of urine. During gestation, hormonal and mechanical factors favor the incidence of urinary loss that may persist after delivery in up to 50% of women. Gestational urine loss can be prevented or treated during pregnancy with physical therapy. Pregnancy and delivery have been widely deemed important risk factors that should be assessed while developing preventive and curative treatments for both female urinary incontinence and pelvic floor muscle dysfunction. Pelvic floor muscle exercises, led by skilled physical therapists, can prevent, reduce, or even cure involuntary urine loss as well as pelvic floor muscle dysfunction. Within this framework, developing a low-cost, easy-to-perform method for the treatment of urinary incontinence and pelvic floor muscle dysfunction, with a preventive or curative approach, is considered necessary. The overall objective of this study is to assess the effects of pelvic floor exercises during pregnancy on pelvic floor muscles and urinary continence. Secondary aims include determining whether exercises change pelvic floor muscle function; if changing pelvic floor muscle function reduces the occurrence of urinary incontinence; developing and applying a manual guide; and determining whether the physical therapy guide is well accepted, easily understandable and reproducible.

DETAILED DESCRIPTION:
Urinary incontinence is any involuntary loss of urine. During gestation, hormonal and mechanical factors favor the incidence of urinary loss that may persist after delivery in up to 50% of women. Gestational urine loss can be prevented or treated during pregnancy with physical therapy. Pregnancy and delivery have been widely deemed important risk factors that should be assessed while developing preventive and curative treatments for both female urinary incontinence and pelvic floor muscle dysfunction. Pelvic floor muscle exercises, led by skilled physical therapists, can prevent, reduce, or even cure involuntary urine loss as well as pelvic floor muscle dysfunction. Within this framework, developing a low-cost, easy-to-perform method for the treatment of urinary incontinence and pelvic floor muscle dysfunction, with a preventive or curative approach, is considered necessary. The overall objective of this study is to assess the effects of pelvic floor exercises during pregnancy on pelvic floor muscles and urinary continence. Secondary aims include determining whether exercises change pelvic floor muscle function; if changing pelvic floor muscle function reduces the occurrence of urinary incontinence; developing and applying a manual guide; and determining whether the physical therapy guide is well accepted, easily understandable and reproducible. Thus, 58 consenting primipregnants aged between 20 and 35 years, with no experience of urinary loss episodes before gestation will be assessed. They will be allocated into 2 groups: G-I: pregnants for the first time who will receive the physical therapy guide, perform the exercises under the supervision of a physical therapist, and complete an exercise compliance form and a log with information on urinary losses; and G-II: pregnants for the first time who will just complete the urinary loss log without receiving the physical therapy guide and performing the exercises. Meetings with each participant will take place at 6 occasions throughout pregnancy: at 18, 22, 26, 30, 34 and 38 weeks of gestation. At 18 weeks, all participants will be asked to respond to a baseline questionnaire with overall and specific gestational data. They will also be questioned about urine loss episodes over the past 30 days, and whether urine loss started during pregnancy. In addition, they will undergo pelvic floor evaluation by Pelvic Floor Functional Assessment (PFFA), and perineometry with a Portable PerinaStim perineometer. G-I women will be taught perineal contraction and receive an exercise guide for perineal contraction in 4 different positions. These women will be instructed to write down exercise frequency on a compliance form as well as the occurrence of urinary incontinence on a urinary loss log. In all 6 meetings, G-I and G-II participants will be reassessed by PFFA and perineometry, and asked to provide their completed urinary loss logs. G-I participants will also be requested to provide their completed exercise compliance form and once again perform the sequence of exercises included in the guide under the supervision of a physical therapist. During all meetings, the notes made on the exercise compliance form will be checked and later added to the baseline form of each participant. The performance of pelvic floor exercises during gestation is expected to have a positive effect on pelvic floor muscles and urinary continence. Pelvic floor muscle function is expected to improve reducing the occurrence of gestational urinary incontinence. In addition, the physical therapy guide is expected to be well accepted, understandable and reproducible. The results obtained in this study are intended to help clinical practice and open new research lines that may significantly contribute to women's health.

ELIGIBILITY:
Inclusion Criteria:

* 58 consenting pregnant for the first time aged between 20 and 35 years, with no experience of urinary loss episodes before gestation will be assessed.

Exclusion Criteria:

* Women who had more than one previous pregnancy

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
UI reduction | 12 months

SECONDARY OUTCOMES:
Pelvic floor muscle dysfunction reduction | 12 monhs

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Dias, Dr., Principal Investigator — Botucatu Medical School
Locations (1):
- Assis Regional Hospital, Assis, São Paulo, Brazil

REFERENCES:
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735
- [Derived] de Assis LC, Bernardes JM, Barbosa AM, Santini AC, Vianna LS, Dias A. [Effectiveness of an illustrated home exercise guide on promoting urinary continence during pregnancy: a pragmatic randomized clinical trial]. Rev Bras Ginecol Obstet. 2015 Oct;37(10):460-6. doi: 10.1590/SO100-720320150005361. Portuguese. PMID 26465164